CLINICAL TRIAL: NCT04393207
Title: Transverse Abdominis Plane Block Using Liposomal Bupivacaine for Post-operative Cesarean Delivery Analgesia- Walking Towards Recovery
Brief Title: TAP Block Using Liposomal Bupivacaine for Post-cesarean Delivery Analgesia- Walking Towards Recovery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow/low recruitment, unable to recruit
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000027606
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use; Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Dexamethasone; Methylprednisolone; Control Groups; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Bupivacaine) (Active Comparator): Patient will receive intrathecal morphine and TAP block with plain bupivacaine.
  Interventions: Drug: Control group (Bupivacaine)- (BPG)
- Liposomal Bupivacaine (Experimental): Patient will receive intrathecal morphine + TAP block with Liposomal bupivacaine and bupivacaine 0.25%
  Interventions: Drug: Liposomal bupivacaine (LB); Drug: Dexamethasone and methylprednisolone (CG)
- Bupivacaine + dexamethasone and methylprednisolone (Active Comparator): Patient will receive intrathecal morphine + TAP block with only bupivacaine.
  Interventions: Drug: Dexamethasone and methylprednisolone (CG)

INTERVENTIONS:
Drug: Liposomal bupivacaine (LB) — Transverse abdominis plane block will be performed and the neurofascial plane between the internal oblique and the transverse abdominis will be infiltrated with liposomal bupivacaine + bupivacaine or with bupivacaine alone.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Dexamethasone and methylprednisolone (CG) — Transverse abdominis plane block will be performed and the neurofascial plane between the internal oblique and the transverse abdominis will be infiltrated with with bupivacaine alone.
  Other Names: Dexamethasone and methylprednisolone
  Arms: Bupivacaine + dexamethasone and methylprednisolone; Liposomal Bupivacaine
Drug: Control group (Bupivacaine)- (BPG) — Transverse abdominis plane block will be performed with plain bupivacaine
  Other Names: Sensorcaine, Marcaine
  Arms: Control group (Bupivacaine)

SUMMARY:
The TAP block offers analgesia by blocking the sensory nerves of the anterior abdominal wall. The procedure is performed under ultrasound guidance, after identification of the external oblique, internal oblique and transverse abdominis muscle. Medication is injected in the neurofascial plane between the internal oblique and the tranversus abdominis muscle.

Previous studies have demonstrated limited (<24 hour) effect of the block when compared to the use of intrathecal morphine (considered to be the "gold standard" for postoperative analgesia). In a study by McMarrow et al., post-caesarian pain control combinations including TAP blocks with local anesthetic (Bupivacaine) or saline after a spinal anesthetic with or without intrathecal morphine were compared.

At 6 hours the Morphine consumption was slightly reduced in the patients that received both intrathecal morphine and TAP blocks with LA when compared to patients that received spinal saline and TAP with saline. At 24 hours the TAP block conferred no benefit in terms of opioid consumption. Similarly, the study by Lee et al. demonstrated better pain scores for the first 2 hours in patients receiving both intrathecal morphine and a TAP block with ropivacaine. At 24 hours there was no difference in the pain scores for patients that received both intrathecal morphine and TAP blocks.

On the contrary, a more recent study utilizing liposomal bupivacaine has been utilized for TAP blocks for post cesarean delivery analgesia, demonstrating opioid reductions for up to 72 hours. Liposomal bupivacaine is a novel, multivesicular formulation designed for rapid absorption, prolonged release of bupivacaine, and analgesia following a single intra-operative administration into the surgical wound or for TAP blocks.

Current anesthesia practices encourage the use of multimodal analgesia that aim at enhanced recovery after surgery (ERAS). The ERAS model aims to decrease immobility, pain and post-operative ileus. Pain and immobility may be closely related, and the latter has rarely been monitored in the post-operative setting. It is planned to use a research validated fit-bit like device (Actigraph GT3-X) to monitor patient steps (mobility).

DETAILED DESCRIPTION:
This is a double blinded, randomized controlled trial. The study will be composed of 3 groups Group 1- Transverse abdominus plain block with liposomal bupivacaine + bupivacaine (LB) Group 2 - Transverse abdominus plain block with bupivacaine (BP) Group 3 - Control group (standard of care with no TAP)

1. Patients will be asked to participate after meeting their anesthesia team and giving verbal consent to receive spinal anesthesia for their cesarean delivery.
2. A computer-generated, single block randomization scheme will be used to allocate patients to one of the three groups (Control group (bupivacaine) Vs TAP LB group or corticosteroid group).
3. In the OR, a spinal using 10-12 mg bupivacaine 0.75%, 10 mcg Fentanyl and 0.1 mg preservative free intrathecal morphine will be performed. Patients will receive IV acetaminophen 1 gram, before skin incision and ketorolac 30 mg after closure of fascia. All patients will receive the same postoperative analgesia orders, which include Tylenol, Ibuprofen and opioids for breakthrough pain. (standard of care)

   After wound closure a TAP block will be performed according to randomization process as described above.
4. The LB TAP block group will receive bilateral ultrasound guided block utilizing 10 ml of liposomal bupivacaine* and 20 ml of 0.25% bupivacaine. The BP TAP group will receive bilateral ultrasound guided block utilizing 20 ml of 0.25% bupivacaine.(Research procedure)
5. The control group will be approached in the exact same way the TAP block group, that is, the ultrasound would be used to identify the muscle layer, but a covered needle will be used to simulate a TAP block. The randomization and procedure will be handled by a co-investigator not involved in the evaluation or data collection at the stablished time points. Patients will be recruited from 7am-5pm and for elective CD
6. The control group will receive Bupivacaine 25 ml of sensorcaine 0.25% + 5 ml saline flush
7. The corticosteroid group will receive sensorcaince 0.25% -20 ml + 10 mg dexamethasone (0.5 ml) + 40 mg methylprednisolone (1 ml) + 8.5 ml normal saline
8. Patients will be asked to complete the ObsQoR-11 at 24 hours, 48 hours and 72 hours.

All patients in this study will be receiving the standard of care. The current standard of care is spinal anesthesia inclusive of intrathecal morphine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 45 presenting for cesarean delivery
2. ASA-1, ASA-2, ASA-3
3. No allergy to morphine
4. No allergy to bupivacaine
5. Patients with BMI > 45 will be excluded
6. No history of anxiety
7. No recent or chronic opioid use

Exclusion Criteria:

1. Need for Magnesium sulfate therapy
2. Neonatal admission to neonatal intensive care unit
3. Need for additional surgery other than cesarean delivery +/- bilateral tubal ligation (e.g. hysterectomy, cystotomy)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gonzalez, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee AJ, Palte HD, Chehade JM, Arheart KL, Ranasinghe JS, Penning DH. Ultrasound-guided bilateral transversus abdominis plane blocks in conjunction with intrathecal morphine for postcesarean analgesia. J Clin Anesth. 2013 Sep;25(6):475-82. doi: 10.1016/j.jclinane.2013.05.004. Epub 2013 Sep 3. PMID 24012493
- [Background] McMorrow RC, Ni Mhuircheartaigh RJ, Ahmed KA, Aslani A, Ng SC, Conrick-Martin I, Dowling JJ, Gaffney A, Loughrey JP, McCaul CL. Comparison of transversus abdominis plane block vs spinal morphine for pain relief after Caesarean section. Br J Anaesth. 2011 May;106(5):706-12. doi: 10.1093/bja/aer061. PMID 21498494
- [Background] Baker BW, Villadiego LG, Lake YN, Amin Y, Timmins AE, Swaim LS, Ashton DW. Transversus abdominis plane block with liposomal bupivacaine for pain control after cesarean delivery: a retrospective chart review. J Pain Res. 2018 Dec 10;11:3109-3116. doi: 10.2147/JPR.S184279. eCollection 2018. PMID 30573987
- [Background] Jacques V, Vial F, Lerintiu M, Thilly N, Mc Nelis U, Raft J, Bouaziz H. [Enhanced recovery following uncomplicated elective caesarean section in France: a survey of national practice]. Ann Fr Anesth Reanim. 2013 Mar;32(3):142-8. doi: 10.1016/j.annfar.2013.01.016. Epub 2013 Feb 19. French. PMID 23433933
- [Background] Alharbi M, Bauman A, Neubeck L, Gallagher R. Validation of Fitbit-Flex as a measure of free-living physical activity in a community-based phase III cardiac rehabilitation population. Eur J Prev Cardiol. 2016 Sep;23(14):1476-85. doi: 10.1177/2047487316634883. Epub 2016 Feb 23. PMID 26907794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group (Bupivacaine) | Liposomal Bupivacaine | Bupivacaine + Dexamethasone and Methylprednisolone
Started | 24 | 60 | 63
Completed | 24 | 60 | 63
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (Bupivacaine) | Liposomal Bupivacaine | Bupivacaine + Dexamethasone and Methylprednisolone | Total
Number analyzed (Participants) | 24 | 60 | 63 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.13 (5.86) | 33.66 (4.79) | 32.8 (5.02) | 33.23 (5.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 60 | 63 | 147
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 10 | 28
  Not Hispanic or Latino | 17 | 49 | 53 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 9 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 9 | 3 | 15
  White | 15 | 46 | 46 | 107
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 24 | 60 | 63 | 147
Gestation [Mean (Standard Deviation); unit: pregnancies] — Previous number of pregnancies
  pregnancies | 2.83 (1.4) | 2.9 (1.72) | 2.4 (0.93) | 2.71 (1.42)
Gestation age in weeks [Mean (Standard Deviation); unit: weeks] | 53.95 (75) | 38.32 (1.62) | 47.36 (56.07) | 45.02 (48.49)

OUTCOME MEASURES:

1. Primary Outcome: Morphine Milligram Equivalents (MME)
Description: Morphine milligram equivalents
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents
Arm/Group | Control Group (Bupivacaine) | Liposomal Bupivacaine | Bupivacaine + Dexamethasone and Methylprednisolone
Number analyzed (Participants) | 24 | 60 | 63
Morphine milligram equivalents | 5.31 (8.12) | 5.16 (10.16) | 5.06 (9.67)

2. Primary Outcome: Morphine Milligram Equivalents (MME)
Description: Morphine milligram equivalents
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents
Arm/Group | Control Group (Bupivacaine) | Liposomal Bupivacaine | Bupivacaine + Dexamethasone and Methylprednisolone
Number analyzed (Participants) | 24 | 60 | 63
Morphine milligram equivalents | 15.31 (22.93) | 15.55 (23.18) | 16.59 (18.15)

3. Primary Outcome: Morphine Milligram Equivalents (MME)
Description: Morphine milligram equivalents
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents
Arm/Group | Control Group (Bupivacaine) | Liposomal Bupivacaine | Bupivacaine + Dexamethasone and Methylprednisolone
Number analyzed (Participants) | 24 | 60 | 63
Morphine milligram equivalents | 6.56 (14.72) | 7.81 (14.51) | 6.56 (11.16)

4. Secondary Outcome: Self Assessed Recovery Survey Obstetric Quality-of-Recovery Score (ObsQoR-11)
Description: Use of a validated questionnaire to measure recovery after cesarean delivery ObsQoR-11. Total score ranging from 0 to 100, with a higher score indicating a better quality of recovery after a caesarean delivery.
Time Frame: 24 hours, 48 hours, 72 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (Bupivacaine) | Liposomal Bupivacaine | Bupivacaine + Dexamethasone and Methylprednisolone
Number analyzed (Participants) | 24 | 60 | 63
score on a scale
  24 hours | 83 (15.3) | 84 (16.1) | 85.2 (15.6)
  48 hours | 80.8 (16.7) | 87.1 (16.6) | 86.6 (15.5)
  72 hours | 86 (41.9) | 90.4 (41.5) | 86 (36.7)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Control Group (Bupivacaine) | Liposomal Bupivacaine | Bupivacaine + Dexamethasone and Methylprednisolone
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/60 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 0/24 | 0/60 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT04393207/Prot_SAP_000.pdf